CLINICAL TRIAL: NCT04976829
Title: Evaluating Antibiotic Stewardship and Healthcare-associated Infections Surveillance Assisted by Computer in the University Hospital of Nancy
Brief Title: Evaluating Antibiotic Stewardship Assisted by Computer in the University Hospital of Nancy (MACABAO)
Acronym: MACABAO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI072
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-07

CONDITIONS: Antibiotic; Healthcare Associated Infection
Keywords: Antibiotic stewardship; Healthcare associated infection; Clinical decision support; Interrupted time series; Infection prevention and control; Antibiotic resistance
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult (≥ 18 years) inpatients (hospitalised ≥ 48h)
  Interventions: Device: Antibiotic stewardship and healthcare-associated infections surveillance assisted by computer

INTERVENTIONS:
Device: Antibiotic stewardship and healthcare-associated infections surveillance assisted by computer — Implementation - in our tertiary care university hospital - of a computerized-decision support system (CDSS) facilitating antibiotic stewardship and of an electronic surveillance software (ESS) facilitating infection prevention and control activities

SUMMARY:
Antibiotic resistance is one of the most pressing health threats that mankind faces now and in the coming decades. Antibiotic resistance leads to longer hospital stays, higher medical costs and increased mortality. In order to tackle antibiotic resistance, a computerized-decision support system (CDSS) facilitating antibiotic stewardship and an electronic surveillance software (ESS) facilitating infection prevention and control activities will implement in our tertiary care university hospital.

The investigators conduct a pragmatic, prospective, single-centre, before-after uncontrolled study with an interrupted time-series analysis 12 months before and 12 months after the introduction of the CDSS for antibiotic stewardship (APSS) and ESS for infection surveillance (ZINC). APSS and ZINC will assist respectively the antibiotic stewardship and the infection prevention and control teams of Nancy University Hospital (France). The investigators will evaluate the impact of the CDSS/ESS on the antibiotic use in adult (≥ 18 years) inpatients (hospitalised ≥ 48h). The primary outcome is the prescription rate by all healthcare professionals from the hospital of all systemic antibiotics expressed in defined daily doses/1 000 patients/month. Concurrently, the investigators will assess the safety of the intervention, its impact on the appropriateness of antibiotic prescriptions and on additional precautions (isolation precautions) as recommended in guidelines, and on bacterial epidemiology (multidrug-resistant bacteria and Clostridioides difficile infections) in the hospital. Finally, the investigators will evaluate the users' satisfaction and the cost of this intervention from the hospital perspective.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients ≥ 18 years and hospitalised ≥ 48h in Nancy University Hospital

Exclusion Criteria:

* The paediatric and gynaeco-obstetric departments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nancy University Hospital (France) is a 1 497-bed tertiary-care hospital including two main geographical sites. In 2017, the point prevalence on one single day of patients treated with antibiotics was 24.4% and the prevalence of HCAI was 7.8% in this University Hospital. And the total antibiotic consumption was 591 DDD/1 000 hospital days.
  The study includes the inpatients of hospital departments of medicine (intensive care, cardiology, hepato-gastro-enterology, haematology, pneumology, infectious diseases, neurology, …), surgery, long-term care, and rehabilitation care.
  All inpatients ≥ 18 years and hospitalised ≥ 48h in Nancy University Hospital will be considered in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Prescription rate of all systemic antibiotics | Calculated monthly during a 12-month before and 12-month after period
  The prescription rate by all healthcare professionals from the Nancy University Hospital of all systemic antibiotics (J01 code according to the Anatomical Therapeutic Chemical - ATC - 2017 classification) expressed in DDDs/1 000 patients/month.

SECONDARY OUTCOMES:
All-cause intra-hospital mortality rate | Calculated monthly during a 12-month before and 12-month after period
  All causes of death/1 000 inpatients/month
Average length of stay | Calculated monthly during a 12-month before and 12-month after period
  Total length of stay for each inpatient/number of stays/month
Incidence of healthcare associated infections | Calculated monthly during a 12-month before and 12-month after period
  New cases of HCAI/ number of inpatients/month
Use of overall antibiotics and by therapeutic classes | Calculated monthly during a 12-month before and 12-month after period
  DDDs/1 000 patients/month
Proportion of the antibiotic prescriptions compliant with guidelines | Calculated monthly during a 12-month before and 12-month after period
  Number of antibiotic prescriptions compliant with guidelines/number of antibiotic prescriptions evaluated
Proportion of the additional precaution prescriptions compliant with hospital recommendations | Calculated monthly during a 12-month before and 12-month after period
  Number of additional precaution prescriptions compliant with hospital recommendations/number of additional precaution prescriptions evaluated
Proportion of C. difficile infections | Calculated monthly during a 12-month before and 12-month after period
  Number of stays with C. difficile infections/number of stays with antibiotic treatment/month
Proportion of multidrug resistant bacteria identification | Calculated monthly during a 12-month before and 12-month after period
  Number of stays with MDRB identification by bacterial sample done after 48h of hospitalization/number of stays with identification of bacterial isolates/month
Hospital costs | During the 12-month after period
  * Costs of antibiotics (costs (in €) of all oral and intravenous antibiotics delivered by hospital pharmacy/month)
  * Average cost of hospital stays (costs (in €) of hospital stays for each inpatient/number of stays/month)
  * Costs of the implementation of the CDSS/ESS and of the purchased equipment (costs (in €) of installation and maintenance of the CDSS/ESS after 12 months of implementation)
Users' satisfaction and acceptability | During the 12-month after period
  * Satisfaction (qualitative study after 6 months of use)
  * Proportion of APSS' alerts accepted by the AMS team (number of APSS' alerts accepted by the AMS team/number of alerts generated by APSS/month)
  * Proportion of AMS team's recommendations accepted by prescribers (number of AMS team's recommendations accepted by prescribers/number of recommendations given by the AMS team to prescribers/month)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Florentin, Dr, Principal Investigator — Université de Lorraine, CHRU-Nancy, APEMAC EA4360, F-54000 Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baudet A, Agrinier N, Charmillon A, Pulcini C, Lozniewski A, Aissa N, Lizon J, Thilly N, Demore B, Florentin A. Evaluating antibiotic stewardship and healthcare-associated infections surveillance assisted by computer: protocol for an interrupted time series study. BMJ Open. 2022 Apr 5;12(4):e056125. doi: 10.1136/bmjopen-2021-056125. PMID 35383069